CLINICAL TRIAL: NCT06769893
Title: A Prospective, Open-label, Single-center Study of CD70-Specific PET/CT Imaging for Non-invasive Diagnosis of Renal Cell Carcinoma
Brief Title: A Study Evaluating the Value of 68Ga-NOTA-RCCB6 PET Imaging for Targeting CD70 in the Clinical Staging, Therapeutic Evaluation, and Restaging of Renal Cell Carcinoma, and Comparing It with 68Ga-PSMA PET/CT Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20242101-F-1; CHiCTR2400084782 (Other: Chinese Clinical Trial Registry)
Record Dates: First submitted 2024-12-22; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: RCC, Renal Cell Cancer
Keywords: Renal cell cancer; PSMA; The cluster of differentiation (CD70); Kidney tumor; ImmunoPET
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: before-after study in the same patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- before-after study in the same patient (Experimental): This is a prospective, open-label, single-center clinical study for renal cell carcinoma.
  Sixty patients clinically suspected of having renal cell carcinoma and undergoing 68Ga-PSMA PET scans were included.
  Qualified subjects underwent 68Ga-NOTA-RCCB6 PET scans within 7 days after completing the 68Ga-PSMA PET scan. Patient medical history was collected and laboratory tests were performed before the examination, and a biopsy or surgery was performed to obtain pathological results within 1 month after the examination, followed by a 6-month follow-up. The pathological results were used as the diagnostic gold standard.
  Interventions: Diagnostic Test: 68Ga-NOTA-RCCB6 PET/CT Scan

INTERVENTIONS:
Diagnostic Test: 68Ga-NOTA-RCCB6 PET/CT Scan — The imaging agent 68Ga-NOTA-RCCB6 used in this project is synthesized following the standards for radiopharmaceutical production, with reference to the Chinese Pharmacopoeia (quality standards for 18F-FDG). The pH value is between 5.0 and 8.0; the radiochemical purity is not less than 95%, and the bacterial endotoxin content in each milliliter of solution is less than 15EU; the radioactive concentration is not less than 37 MBq/mL; the solvent residues comply with the regulations.
  Specification: 185~1850 MBq/ml Characteristics: Clear, colorless, no visible particles. Radioactive physical half-life: 68Ga is 68 minutes. Expiry: Calculated from the time of labeling, stable for 3 half-lives. Administration method: Intravenous injection. Dosage: 0.05-0.1mCi/kg, flush with 5 mL of saline after injection. The maximum mass dose of CD70 should not exceed 240ug, and the maximum volume of administration should not exceed 5 mL.

SUMMARY:
This is a prospective, open-label, single-center clinical study targeting renal cell carcinoma. Sixty patients with a high clinical suspicion of renal cell carcinoma were included. Qualified subjects will undergo 68Ga-NOTA-RCCB6 PET/CT examination. The aim is to establish the optimal imaging protocol; evaluate the distribution characteristics and correlations of physiological and pathological positive uptake, and using pathological results as the gold standard, assess the diagnostic efficacy of 68Ga-NOTA-RCCB6 PET/CT in renal cell carcinoma.

DETAILED DESCRIPTION:
This research process is divided into screening period, baseline period, safety visit period, and diagnostic efficacy follow-up period.

1. Screening period (D-7 to D-1): No more than 7 days

   Screening is conducted within 7 days before the administration of 68Ga-NOTA-RCCB6 (D-7 to D-1). Before any study-related procedures, subjects must sign a written informed consent form. After signing the informed consent form, the following screening procedures are performed:

   ① Review of inclusion/exclusion criteria.
   * Collection of medical history, including but not limited to clinical data of the subjects and relevant auxiliary examination results (routine imaging examinations, tumor markers, biopsy results, etc.), numbering each subject and establishing a medical record.

     * Collection of demographic data (including gender, age, etc.). ④ Recording of concomitant medications/adverse events. If any inclusion criteria are not met or any exclusion criteria are met, the screening is considered failed.
2. Baseline period (drug/administration period) (D0): 1 day Subjects who meet all inclusion criteria and do not meet any exclusion criteria will receive an injection of 68Ga-NOTA-RCCB6 and undergo a PET/CT scan on D0. The following assessments are performed again before administration, and only after a comprehensive evaluation by the doctor are they eligible for injection.

   * Concomitant medications after screening visit ② Weight

     * Vital signs

       * Adverse events Single dose, 0.05-0.1mCi/kg body weight, intravenous injection of 68Ga-NOTA-RCCB6 0.05-0.1mCi/kg PET/CT scan is performed 50-80 minutes after administration.
3. Safety visit period (D0 to D4): 4 days

   * Follow-up on whether subjects have adverse reactions after administration.

     ② 2 hours ± 10 minutes after administration: monitoring of adverse events in subjects.

     ③ 1-4 days after administration: telephone follow-up to assess for delayed adverse events.
4. Diagnostic efficacy follow-up period (D1 to D180): 6 months Follow-up on biopsy/surgical pathology results of subjects (preferably completed within 1 month after imaging) and imaging results to confirm the diagnostic efficacy of 68Ga-NOTA-RCCB6 PET/CT in renal cell carcinoma.

   When conducting diagnostic efficacy follow-up, the following should be recorded simultaneously: concomitant medications and adverse events.
5. Withdrawal from study/premature termination of study

   If patients do not complete the PET examination according to the process, for subjects who withdraw prematurely, the following follow-up should be completed:

   ① Concomitant medications

   ② Adverse events
6. Premature termination or suspension of study Reasons for study termination may include but are not limited to: new information on safety, requirements of the competent authorities. Other reasons include but are not limited to: excessive protocol violations, insufficient concern for subject safety, researcher turnover or insufficient staffing, etc.

In the event of any of the following situations during the study, the study may be terminated, and the competent authority should promptly report to the health department responsible for clinical research registration:

* There is a violation of laws and regulations, rules;

  * There is a violation of ethical principles or the principles of scientific integrity;

    * During the study, it is found that the study drug may have serious quality defects; ④ Serious safety risks are found in clinical research;

      * There is commercial bribery or other improper interest relationships; ⑥ Other situations that should stop the study. For all situations where the study is suspended or terminated, appropriate steps will be taken to ensure the safety of the subjects.

Definition of study completion: PET imaging, result analysis, and necessary clinical follow-up of all study subjects have been completed.

ELIGIBILITY:
Inclusion Criteria:

- The subject or legal guardian/caregiver must voluntarily sign the informed consent form.

Ages 18 to 75 years old. Patients with suspected renal cell carcinoma based on conventional imaging studies, and who undergo 68Ga-PSMA PET/CT scanning.

Patients with suspicious lymph nodes or distant metastases detected by conventional imaging or 68Ga-PSMA PET/CT.

Willing and able to follow the study protocol.

Exclusion Criteria:

- Patients who have received anti-tumor treatment prior to PET/CT scan. Suffer from severe other neurological diseases, or gastrointestinal, cardiovascular, liver, kidney, blood system, respiratory system, immunodeficiency and other serious diseases.

Alternative subjects have contraindications to PET/CT scanning. Including but not limited to: those who cannot tolerate repeated intravenous injections; those who may be allergic to the drug and its components (including those with a history of severe allergies or allergic reactions, especially those with allergies to the tested drug); claustrophobia.

In the past year, diagnosed with other malignant tumors; alternative subjects have undergone major surgery in the past 3 months; received experimental drug or device treatment with unclear effects or safety within the past month, or have participated in other interventional clinical trials.

Pregnant or lactating women. Patients who are lost to follow-up. Other conditions that, in the researcher's assessment, may affect the study or make the subject unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-11-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Standardized uptake value (SUVmax) | 1 day from injection of the tracer
  Maximum Standardized uptake value (SUVmax) of [68Ga]RCCB6 and [68Ga]PSMA in the included subjects' primary and/or metastatic lesions.
Mean Standardized Uptake Value(SUVmean) of liver | 1 day from injection of the tracer
  Mean Standardized uptake value (SUVmean) of [68Ga]RCCB6 and [68Ga]PSMA in the included subjects' liver.
Tumor to Background Ratio(TBR) | 1 day from injection of the tracer
  TBR=SUVmax/SUVmean
The correlation between CD70 expression and [18F]RCCB6 uptake value | 30 days from injection of the tracer
  The Standardized uptake value (SUV) of [68Ga]RCCB6 will be calculated, and the correlation between pathological results and tumor uptake of [68Ga]RCCB6 will be analyzed.

SECONDARY OUTCOMES:
Diagnostic value of 68Ga-NOTA-RCCB6 PET/CT in patients with RCC | 3-6 months from injection of the tracer
  We will calculate the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy of 68Ga-NOTA-RCCB6 PET/CT in patients with RCC. We will also compare the diagnostic value of [68Ga]RCCB6 with [68Ga]PSMA. All the above goals will be achieved by analyzing the 68Ga-NOTA-RCCB6 PET/CT and 68Ga-PSMA PET/CT imaging data.

CONTACTS AND LOCATIONS:
Locations (1):
- Department ofNuclear Medicine,Xijing Hospital, Fourth Military Medical University, Xi'an, China, Xi'an, China, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ChiCTR2400084782 registration number of the Chinese Clinical Trial Registry — http://www.medresman.org.cn